CLINICAL TRIAL: NCT05946213
Title: The Phase III 'High Five Trial' Five Fraction Radiation For High-Risk Prostate Cancer
Brief Title: Testing Shorter Duration Radiation Therapy Versus the Usual Radiation Therapy in Patients With High Risk Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU013; NCI-2023-04142 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU013 (Other: NRG Oncology); NRG-GU013 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2023-06-28; First posted 2023-07-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostate Adenocarcinoma; Stage III Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Congresses as Topic; Radiation; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (SBRT) (Experimental): Patients undergo SBRT for a total of 5 treatments over 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo bone scan and/or CT, MRI, or PET/CT during screening and CT and/or MRI on study. Additionally, patients may optionally undergo blood and urine sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy
- Arm II (EBRT) (Active Comparator): Patients undergo EBRT for 20 to 45 treatments over 4 to 9 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo bone scan and/or CT, MRI, or PET/CT during screening and CT and/or MRI on study. Additionally, patients may optionally undergo blood and urine sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
  Arms: Arm I (SBRT)
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
  Arms: Arm II (EBRT)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Arm I (SBRT)

SUMMARY:
This phase III trial compares stereotactic body radiation therapy (SBRT), (five treatments over two weeks using a higher dose per treatment) to usual radiation therapy (20 to 45 treatments over 4 to 9 weeks) for the treatment of high-risk prostate cancer. SBRT uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period of time. This trial is evaluating if shorter duration radiation prevents cancer from coming back as well as the usual radiation treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare metastasis-free survival, determined using conventional imaging, between men with high-risk prostate cancer randomized to ultrahypofractionation (stereotactic body radiation therapy [SBRT]) to those randomized to moderate hypofractionation and conventional fractionation.

SECONDARY OBJECTIVES:

I. To compare physician-reported toxicity as measured by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5 between treatment arms.

II. To determine if ultrahypofractionation is non-inferior to moderate hypofractionation and conventional fractionation with respect to patient-reported urinary function (assessed by Expanded Prostate Cancer Index Composite [EPIC]-26 urinary domains).

III. To determine if ultrahypofractionation is non-inferior to moderate hypofractionation and conventional fractionation with respect to patient-reported bowel function (assessed by EPIC-26 bowel domain).

IV. To compare patient-reported fatigue (assessed by Patient Reported Outcomes Measurement Information System [PROMIS]-Fatigue) between treatment arms.

V. To compare failure-free survival between treatment arms. VI. To compare metastasis-free survival based on molecular imaging between treatment arms.

VII. To compare overall survival between treatment arms.

EXPLORATORY OBJECTIVES:

I. To compare patient-reported sexual function (assessed by EPIC-26 sexual domain) between treatment arms.

II. To compare patient-reported quality of life (assessed by European Quality of Life Five Dimension Five Level Scale Questionnaire [EQ-5D-5L]) between treatment arms.

III. To compare patient-reported treatment burden (assessed by COmprehensive Score for financial Toxicity (COST)) between treatment arms

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo SBRT for a total of 5 treatments over 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo bone scan and/or computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET)/CT during screening and CT and/or MRI on study. Additionally, patients may optionally undergo blood and urine sample collection on study.

ARM II: Patients undergo external beam radiation treatment (EBRT) for 20-45 treatments over 4 to 9 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo bone scan and/or CT, MRI, or PET/CT during screening and CT and/or MRI on study. Additionally, patients may optionally undergo blood and urine sample collection on study.

Patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of adenocarcinoma of prostate cancer
* High-risk disease defined as having at least one or more of the following:

  * cT3a-T3b by digital exam or imaging (American Joint Committee on Cancer [AJCC] 8th edition [Ed.]) Note: cT4 by imaging or on digital rectal exam is not allowed
  * The patient's prostate specific antigen (PSA) value > 20 ng/mL prior to starting androgen deprivation therapy (ADT) Note: Patients taking a 5-alpha reductase inhibitor (ex finasteride or dutasteride) are eligible The baseline PSA value should be doubled for PSAs taken while on 5-alpha reductase inhibitors
  * Gleason Score of 8-10
  * Pelvic node positive by conventional imaging with a short axis of at least 1.0 cm
* Prostate gland volume less than 100 cc prior to initiation of ADT as reported at time of biopsy or by separate measure with ultrasound or other imaging modalities including MRI or CT scan
* No definitive clinical or radiologic evidence of metastatic disease outside of the pelvic nodes (M1a, M1b or M1c) on conventional imaging (i.e. bone scan, CT scan, MRI); Negative prostate-specific membrane antigen (PSMA) positron emission tomography (PET) is an acceptable substitute
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* No prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* No prior radical prostatectomy
* No prior ablative or focal therapy to the prostate (including, but not limited to, transrectal or transurethral high-intensity focused ultrasound [HIFU], laser ablation, cryotherapy, irreversible electroporation [IRE], and vascular-targeted photodynamic therapy)
* Prior pharmacologic androgen ablation for prostate cancer is allowed only if the onset of androgen ablation (both luteinizing hormone releasing hormone [LHRH] agonist and oral anti-androgen) is =< 185 days prior to registration; Please note: PSA prior to the start of any ADT will be used to define disease
* No contraindication to prostate MRI (required for planning of radiotherapy in both arms)
* Patients enrolled in NRG-GU009 must be enrolled in NRG-GU013 prior to radiation therapy treatment planning and start of radiation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1209 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2036-03-31 (Estimated); Study Completion 2036-03-31 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival (MFS) | From randomization to the date of distant metastasis, or death from any cause, assessed up to 15 years
  Based on conventional imaging. Median MFS time comparing the curves.

SECONDARY OUTCOMES:
Failure-free survival | From randomization to the date of distant metastasis, or death from any cause, assessed up to 15 years
  Median failure-free survival time comparing the curves.
Overall survival | From the date of randomization to the date of death or last known follow-up date, with patients alive at the last known follow-up time treated as censored, assessed up to 15 years
  Median survival time comparing the curves.
MFS | From randomization to the date of distant metastasis, or death from any cause, assessed up to 15 years
  Median MFS time comparing the curves.
Incidence of adverse events (AEs) | Up to 15 years
  AEs will be graded using National Cancer Institute's (NCI's) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5. Counts of all AEs by grade will be provided by treatment arm.
Urinary incontinence | Up to 5 years
  Proportion of patients with a decline, as measured by the urinary incontinence domain of the Expanded Prostate Cancer Index Composite (EPIC-26).
Urinary irritative/obstructive | Up to 5 years
  Proportion of patients with a decline, as measured by the urinary irritative/obstructive domain of the Expanded Prostate Cancer Index Composite (EPIC-26).
Bowel function | Up to 5 years
  Proportion of patients with a decline, as measured by the bowel domain of the Expanded Prostate Cancer Index Composite (EPIC-26).
Fatigue | Up to 5 years
  Proportion of patients with a decline, as measured by the Patient Reported Outcomes Measurement Information System-Fatigue.

OTHER OUTCOMES:
Patient-reported outcomes | Up to 5 years
  The EPIC-26 sexual domain will be assessed as an exploratory endpoint but following the analysis plan specified for the EPIC-26 urinary and bowel domains.
Cost | Up to 1 year
  Measured by the Functional Assessment of Chronic Illness Therapy-COST.
Estimate of treatment effect by sex | Up to 15 years
  Will estimate the primary outcome treatment effect and the corresponding 95% confidence intervals (CIs) by sex.
Estimate of treatment effect by race | Up to 15 years
  Will estimate the primary outcome treatment effect and the corresponding 95% CIs by race.
Estimate of treatment effect by ethnicity | Up to 15 years
  Will estimate the primary outcome treatment effect and the corresponding 95% CIs by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Hoffman, Principal Investigator — NRG Oncology
Locations (383):
- United States (373):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Lewis and Faye Manderson Cancer Center, Tuscaloosa, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Moffitt Cancer Center at SouthShore, Ruskin, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Alton Memorial Hospital, Alton, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Gonzales, Gonzales, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Veterans Administration Medical Center-Baltimore, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - UM Capital Region Medical Center, Largo, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Jersey City Medical Center, Jersey City, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Sands Cancer Center, Canandaigua, New York
  - Noyes Memorial Hospital/Myers Cancer Center, Dansville, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Northwell Health Physicians Partners Radiation Medicine at Queens, Forest Hills, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - Upstate Cancer Center Radiation Oncology at Oswego, Oswego, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Upstate Cancer Center at Hill Radiation Oncology, Syracuse, New York
  - Westchester Medical Center, Valhalla, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Durham VA Medical Center, Durham, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - MD Anderson in The Woodlands, Conroe, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - VCU Massey Cancer Center at Hanover Medical Park, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (8):
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- Kantonsspital Aarau, Aarau, Switzerland